CLINICAL TRIAL: NCT00638885
Title: Memory and the Hippocampus in Vietnam Twins With PTSD
Brief Title: Memory and the Hippocampus in Twins
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: MHBA-008-07S
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Results first posted 2015-01-15 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: PTSD; Stress Disorders, Post-Traumatic
Keywords: PTSD; hippocampus; twins
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood for genetic testing, blood samples and urine and saliva collections
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
The purpose of this project is to measure brain markers and cognitive factors in twins with a history of military service with and without PTSD, and to follow them over time and measure changes in brain function and cognitive variables.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a condition of critical importance to the Veterans Health Administration that affects up to 15% of Vietnam combat veterans.1 Studies in animals demonstrated that stress is associated with alterations in the morphology of the hippocampus, a brain structure involved in learning and memory, as well as memory deficits. Patients with PTSD have smaller hippocampal volume on magnetic resonance imaging (MRI) and deficits in memory on neuropsychological testing. Animal models also show a progressive diminution of hippocampal volume with normal aging that is associated with a loss of memory function. In humans, in very old age in some individuals the hippocampus becomes smaller, with associated declines in memory function. Clinically, PTSD patients appear to have a more rapid rate of memory decline with age, which has led to their being characterized as having an "accelerated aging"; however there is little empiric data related to the interaction between normal aging and PTSD and its effect on memory. In the prior period of VA Merit funding the PI has studied memory and the hippocampus in twin pairs discordant for PTSD as well as normal twin pairs. We have studied 42 MZ and DZ twin pairs discordant for Vietnam theater exposure and discordant for PTSD and 28 MZ and DZ twin pairs concordant for Vietnam theater exposure and discordant for PTSD. All twins underwent measures of hippocampal volume, neuropsychological testing, and cortisol. A subset of 10 pairs of MZ pairs discordant for PTSD and combat exposure underwent positron emission tomography (PET) imaging of neural correlates of declarative memory function. Preliminary analyses are consistent with smaller hippocampal volume and deficits in verbal declarative memory in PTSD affected twins compared to their non-PTSD brothers who were not exposed to Vietnam combat.

We now propose to measure hippocampal volume, memory function, and neural correlates of declarative memory, in MZ and DZ twins previously studied, who are discordant for combat and PTSD. We will study 42 twin pairs who were studied during 1999-2003, of whom 34 were discordant for PTSD at the Atlanta based assessment and had all study data including MRI, neuropsychological testing, and cortisol (with PET in a subsample of 10 pairs), with repeat measurements performed 8 years after the initial assessment, a time of life when they become vulnerable to memory decline associated with aging (subjects not discordant for PTSD at the Atlanta based assessment will also be studied as a comparison). These assessments will allow a comprehensive assessment of the relative impact of shared environment (e.g. family life), unique environment (Vietnam theater service), and genetics on the outcomes of interest. We hypothesize that there will be an interaction between PTSD diagnosis and aging, i.e. PTSD patients relative to non-PTSD will show smaller hippocampal volume as measured with MRI, deficits in verbal declarative memory as measured with neuropsychological testing, lower cortisol, and a failure of hippocampal function during memory tasks as measured with PET, and that the rate of decline will be greater in PTSD v non PTSD. We further hypothesize that analysis of all twin pair combinations will show a combined impact of genetics and PTSD diagnosis on the hippocampal outcomes of interest.

ELIGIBILITY:
Inclusion Criteria:

* All twins will be required to give written informed consent.
* Subjects will be included with a history of Vietnam Era service.
* All subjects must be free of major medical illness on the basis of history and physical examination, lab testing, and electrocardiogram.

Exclusion Criteria:

* Subjects will be excluded with a history of shrapnel or other foreign bodies that would preclude MRI scanning, history of loss of consciousness, or neuroleptics, sedative or benzodiazepine medication usage within the previous four weeks.
* Subjects will also be excluded if based on the SCID interview they have comorbid:

  * schizophrenia;
  * schizoaffective disorder;
  * bulimia or anorexia, or
  * bipolar disorder.
* Subjects will also be excluded with a history of blast injury with associated traumatic brain injury.
* In addition, subjects will be excluded with a history of alcohol or substance abuse/dependence within the past year. We will use the strategy used in prior MRI studies and use multivariate analyses to examine the contribution of past histories of alcohol and substance abuse (as measured with the Addiction Severity Index) and depression symptom level (as measured with the Hamilton Depression Scale) to the outcomes of interest.
* Subjects will be excluded from the study if they present with a history of serious medical or neurological illness, or as a result of routine laboratory studies, history of asthma, steroid usage, seizure disorder, or prenatal/perinatal substance exposure or trauma.

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twins with history of military service during Vietnam era with and without PTSD
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2010-04; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doug Bremner, MD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia, United States

REFERENCES:
- See also: J. Douglas Bremner, M.D. Website — http://www.dougbremner.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited through Vietnam Era Twin Registry 2001-2012.
Pre-assignment Details: Subjects studied at baseline with no interventions.
Groups:
- Group 1: Vietnam veterans who were twins with and without posttraumatic stress disorder underwent neuropsychological testing and MRI imaging of hippocampal volume at baseline. There were no clinical interventions.
Period: Overall Study
Arm/Group | Group 1
Started | 142
Completed | 142
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Vietnam veteran twins with and without PTSD.
Arm/Group | Group 1
Number analyzed (Participants) | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 142
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 142
Region of Enrollment [Number; unit: participants]
  United States | 142

OUTCOME MEASURES:

1. Primary Outcome: Neuropsychological Testing of Memory
Description: Percent retention on the Wechsler Memory Scale - Logical
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: percentage of WMS retention
Groups:
- Vietnam Veteran Twins: Vietnam veteran twins with and without PTSD.
Arm/Group | Vietnam Veteran Twins
Number analyzed (Participants) | 142
percentage of WMS retention
  PTSD | 77 (14)
  non PTSD | 82 (15)

ADVERSE EVENTS:
Arm/Group | Vietnam Twins With and Without PTSD
Serious Adverse Events (participants affected / at risk) | 0/142
Other Adverse Events (participants affected / at risk) | 0/142

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes